CLINICAL TRIAL: NCT05740059
Title: Restrictive Transfusion StratEgy Adjusted by SvO2 During Cardiac Surgery: Multicenter, Single-blinded, Randomised Controlled Trial.
Brief Title: Restrictive Transfusion StratEgy Adjusted by SvO2 During Cardiac Surgery
Acronym: RETSEACSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL21_0529
Record Dates: First submitted 2023-02-06; First posted 2023-02-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Blood transfusion; Cardiac surgery

STUDY DESIGN:
Intervention Model Description: Multi-center, single-blinded, and randomized controlled trial.
Who Masked: Participant
Masking Description: Patients won't be aware of the assignment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients assigned to the Control group will be transfused if hemoglobin (Hb) concentration is lower than 9 g/d.
- Adjusted transfusion (Active Comparator): Patients assigned to the SvO2 group will be transfused if Hb concentration is lower than 9 g/dL and central SvO2 ≤ 65%.
  Interventions: Other: Adjusted Transfusion

INTERVENTIONS:
Other: Adjusted Transfusion — Patients assigned to the SvO2 group will be transfused if Hb concentration is lower than 9 g/dL and central SvO2 ≤ 65%. Transfusion will be repeated whenever Hb concentration is lower than 9 g/dL and central SvO2 ≤ 65% during surgery and in the ICU (until day 5). Central SvO2 will be measured on a blood sample obtained from the distal lumen of the central venous catheter. Oximetry will be used for measurement with a point-of-care of gas analysis.
  Arms: Adjusted transfusion

SUMMARY:
The goal of the clinical trial is to evaluate whether a restrictive transfusion strategy adjusted by SvO2 during the perioperative period of cardiac surgery may reduce the incidence of red blood cell transfusion. Adult patients operated on cardiac surgery will be randomly allocated into two groups, one receiving standard restrictive transfusion, the other receiving SvO2 adjusted restrictive transfusion.The proportion of patients transfused will be compared between the 2 groups.

DETAILED DESCRIPTION:
Cardiac surgery represents only a small fraction of all surgical procedures, but consumes a significant proportion of the stored red blood cells (RBC), with almost 50% of patients receiving a perioperative transfusion. Since RBC transfusion is associated with an increased risk of morbidity and mortality, blood patient management strategy has been promoted to favour prevention of anaemia, reduction of bleeding and limitation of transfusion. Current guidelines recommend haemoglobin (Hb) threshold as low as 7 g/dL, but still with a wide possible range (7 to 9 g/dl) and suggest that Hb alone may not be the best criteria for triggering transfusion. As Hb is an oxygen carrier, the rationale for RBC transfusion should be to increase tissue oxygen delivery. Central venous oxygen saturation (central SvO2), which is related to the balance between tissue oxygen delivery and consumption, is easily measurable in cardiac surgery. In a previous study, the investigators showed that in anaemic patients having undergone cardiac surgery, restrictive transfusion according to central SvO2 allowed a significant reduction in RBC transfusion incidence in the ICU. The investigators hypothesize that a restrictive transfusion strategy adjusted by SvO2 during all the perioperative period of cardiac surgery may reduce further the incidence of RBC transfusion. Limiting RBC transfusion to patients with a low SvO2 could save unnecessary transfusions, without increasing the anaemia related risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years and under 85 years
* Signed informed consent form from the patient or his/her close relative or surrogate (if present) before inclusion or when possible when the patient has been included in an emergency setting
* Anaemic (Haemoglobin at inclusion ≤ 13 g/dL)
* Operated on elective, on-pump cardiac surgery for : Coronary artery bypass graft (CABG); Aortic, mitral or tricuspid valve (replacement or repair); Ascending aorta;Left ventricle assistance device (LVAD)
* Operated on urgent on-pump cardiac surgery for : CABG;Endocarditis;Aortic dissection; Heart transplantation
* Subjects must be covered by public health insurance

Exclusion Criteria:

* Patient with no central venous catheter inserted in the superior vena cava
* Pregnant or breast feeding patient
* Subject unable to read or/and write
* Participation in another interventional clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date
* Medical history of heparin-induced thrombocytopenia contraindicating heparin use during surgery
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric care and persons admitted to a health or social establishment for purposes other than research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
RBC transfusion incidence | During cardiac surgery and postoperative ICU stay up to postoperative day 5
  Proportion of RBC transfused patients

SECONDARY OUTCOMES:
RBC transfusion incidence during surgery | During cardiac surgery
  Proportion of patients transfused with RBC during surgery
RBC units transfused during surgery | During cardiac surgery
  Number of RBC units transfused during surgery
RBC transfusion incidence during postoperative ICU stay | During postoperative ICU stay
  Proportions of patients transfused with RBC during postoperative ICU stay
RBC units transfused during postoperative ICU stay | During postoperative ICU stay
  Number of RBC units transfused during postoperative stay in ICU
RBC transfusion incidence at hospital discharge or day 28 | From cadiac surgery to hospital discharge or day 28
  Proportions of patients transfused with RBC at hospital discharge or day 28
RBC units transfused at hospital discharge or day 28 | From cardiac surgery to hospital discharge or day 28
  Number of RBC units transfused at hospital discharge or day 28
Postoperative septic complications | From cardiac surgery to hospital discharge or day 28
  Proportion of postoperative septic complications
Postoperative ischemic complications | From cardiac surgery to hospital discharge or day 28
  Proportion of postoperative ischemic complications (myocardial infarction, stroke, mesenteric)
Postoperative acute kidney injury | From cardiac surgery to hospital discharge or day 28
  Proportion postoperative AKI according to Kdigo stages
Postoperative liver dysfuncion | From cardiac surgery to hospital discharge or day 28
  Proportion of postoperative increase in binirubin or plasma hepatic enzymes
Postoperative respiratory failure | From cardiac surgery to hospital discharge or day 28
  Proportion of postoperative of Pa/Fi<200
Postoperative low cardiac output syndrome | From cardiac surgery to hospital discharge or day 28
  Proportion of low cardiac output
Postoperative arythmias | From cardiac surgery to hospital discharge or day 28
  Proportion of atrial fibrillation
Length of ICU stay | From ICU admission to ICU discharge ofr day 28
  ICU length of stay (number of days)
Length of hospital stay | From ICU admission to hospital discharge or day 28
  Hospital length of stay (number of days)
Postoperative anemia | From ICU admission to hospital discharge or day 28
  Hemoglobin concentration
Death | From cardiac surgery to hospital discharge or day 28
  Proportion of deaths
Effect of RBC transfusion on Hb | During cardiac surgery and postoperative ICU stay up to postoperative day 5
  Hb changes after RBC transfusion
Effect of RBC transfusion on central SvO2 | During cardiac surgery and postoperative ICU stay up to postoperative day 5
  Central SvO2 changes after RBC transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Departement d'anesthésie et réanimation D - Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bennett-Guerrero E, Zhao Y, O'Brien SM, Ferguson TB Jr, Peterson ED, Gammie JS, Song HK. Variation in use of blood transfusion in coronary artery bypass graft surgery. JAMA. 2010 Oct 13;304(14):1568-75. doi: 10.1001/jama.2010.1406. PMID 20940382
- [Result] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Ferraris SP, Saha SP, Hessel EA 2nd, Haan CK, Royston BD, Bridges CR, Higgins RS, Despotis G, Brown JR; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Spiess BD, Shore-Lesserson L, Stafford-Smith M, Mazer CD, Bennett-Guerrero E, Hill SE, Body S. Perioperative blood transfusion and blood conservation in cardiac surgery: the Society of Thoracic Surgeons and The Society of Cardiovascular Anesthesiologists clinical practice guideline. Ann Thorac Surg. 2007 May;83(5 Suppl):S27-86. doi: 10.1016/j.athoracsur.2007.02.099. PMID 17462454
- [Result] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Result] Stover EP, Siegel LC, Parks R, Levin J, Body SC, Maddi R, D'Ambra MN, Mangano DT, Spiess BD. Variability in transfusion practice for coronary artery bypass surgery persists despite national consensus guidelines: a 24-institution study. Institutions of the Multicenter Study of Perioperative Ischemia Research Group. Anesthesiology. 1998 Feb;88(2):327-33. doi: 10.1097/00000542-199802000-00009. PMID 9477051
- [Result] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Result] Koch CG, Li L, Duncan AI, Mihaljevic T, Loop FD, Starr NJ, Blackstone EH. Transfusion in coronary artery bypass grafting is associated with reduced long-term survival. Ann Thorac Surg. 2006 May;81(5):1650-7. doi: 10.1016/j.athoracsur.2005.12.037. PMID 16631651
- [Result] Paone G, Likosky DS, Brewer R, Theurer PF, Bell GF, Cogan CM, Prager RL; Membership of the Michigan Society of Thoracic and Cardiovascular Surgeons. Transfusion of 1 and 2 units of red blood cells is associated with increased morbidity and mortality. Ann Thorac Surg. 2014 Jan;97(1):87-93; discussion 93-4. doi: 10.1016/j.athoracsur.2013.07.020. Epub 2013 Oct 3. PMID 24094521
- [Result] American Society of Anesthesiologists Task Force on Perioperative Blood Management. Practice guidelines for perioperative blood management: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Management*. Anesthesiology. 2015 Feb;122(2):241-75. doi: 10.1097/ALN.0000000000000463. No abstract available. PMID 25545654
- [Result] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- [Result] Pagano D, Milojevic M, Meesters MI, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Boer C. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):79-111. doi: 10.1093/ejcts/ezx325. No abstract available. PMID 29029100
- [Result] Mazer CD, Whitlock RP, Fergusson DA, Hall J, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, McGuinness S, Royse A, Carrier FM, Young PJ, Villar JC, Grocott HP, Seeberger MD, Fremes S, Lellouche F, Syed S, Byrne K, Bagshaw SM, Hwang NC, Mehta C, Painter TW, Royse C, Verma S, Hare GMT, Cohen A, Thorpe KE, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Restrictive or Liberal Red-Cell Transfusion for Cardiac Surgery. N Engl J Med. 2017 Nov 30;377(22):2133-2144. doi: 10.1056/NEJMoa1711818. Epub 2017 Nov 12. PMID 29130845
- [Result] Fominskiy E, Putzu A, Monaco F, Scandroglio AM, Karaskov A, Galas FR, Hajjar LA, Zangrillo A, Landoni G. Liberal transfusion strategy improves survival in perioperative but not in critically ill patients. A meta-analysis of randomised trials. Br J Anaesth. 2015 Oct;115(4):511-9. doi: 10.1093/bja/aev317. PMID 26385661
- [Result] Zeroual N, Blin C, Saour M, David H, Aouinti S, Picot MC, Colson PH, Gaudard P. Restrictive Transfusion Strategy after Cardiac Surgery. Anesthesiology. 2021 Mar 1;134(3):370-380. doi: 10.1097/ALN.0000000000003682. PMID 33475735
- [Result] Colson PH, Gaudard P, Fellahi JL, Bertet H, Faucanie M, Amour J, Blanloeil Y, Lanquetot H, Ouattara A, Picot MC; ARCOTHOVA group. Active Bleeding after Cardiac Surgery: A Prospective Observational Multicenter Study. PLoS One. 2016 Sep 2;11(9):e0162396. doi: 10.1371/journal.pone.0162396. eCollection 2016. PMID 27588817